CLINICAL TRIAL: NCT06179589
Title: Clinical Trial to Compare the Efficacy and Safety of a Multiple Amino-acid Based ORS "VS002A" With the Standard WHO-ORS in the Management of Noncholera Acute Watery Diarrhea in Infants and Young Children
Brief Title: VS002A in the Treatment of Acute Watery Diarrhea in Infants and Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Entrinsic Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-17028
Record Dates: First submitted 2021-02-01; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-04

CONDITIONS: Acute Watery Diarrhoea

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, parallel group, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VS002A (Experimental): Advanced Amino acid-based ORS: VS002A Traditional oral rehydration solutions (ORS) contain sugars which stimulate intestinal sodium and water absorption through a variety of mechanisms. However, it has been under-appreciated that traditional ORS possess no anti-diarrheal functions and may exacerbate infectious diarrheal secretions.
  Interventions: Dietary Supplement: VS002A
- WHO-ORS (Active Comparator): WHO-ORS usually used worldwide in the treatment of diarrhoea.
  Interventions: Dietary Supplement: VS002A

INTERVENTIONS:
Dietary Supplement: VS002A — Amino acid based, glucose free ORS

SUMMARY:
Background (brief):

1. Burden: Diarrhea is the second deadliest disease for under-five children globally and the situation is more serious in developing countries. It was responsible for 688 million illnesses and 499,000 deaths worldwide in children less than 5 years of age in 2015 (Kotloff, 2017). Majority of the deaths from diarrhea occur before the second birthday of the children and it contributes to more than 20% of overall death in infants and young children.
2. Knowledge gap: Oral rehydration solution (ORS) is being used as a standard treatment for acute watery diarrhea for long time and which is one of the best inventions in the history of medicine. The ORS currently recommended by the WHO/UNICEF contains glucose, sodium chloride, potassium chloride, and tri-sodium citrate dehydrate, which is optimal for rehydration of patients of all ages with dehydration from acute diarrhea of any aetiology. However, oral rehydration therapy (ORT) with the present ORS formulation has certain limitations - it does not reduce the volume, frequency or the duration of diarrhea. Additionally, the failure of present standard ORS to reduce dramatically stool output likely contributes to the relatively limited use of ORS by mothers as they do not feel that ORS is helping their child from the episode of diarrhea. Thus, it warrants the development of newer and improved formulation of ORS to become more effective against diarrhea.
3. Relevance: It has been reported that the glucose contained in standard ORS may fail to absorb fluid and electrolytes adequately from gut and worsen diarrhea in different patho-physiological ways as the present WHO ORS is hypo-osmolar. Whereas, certain neutral amino acids (e.g. glycine, L-alanine, L-glutamine) are able to enhance the absorption of sodium ions and water from gut. By using this concept, the University of Florida (UF), developed a sugar-free, shelf-stable amino acid-based hydration medicinal food named 'VS002A' that effectively rehydrates, and improves barrier function of the bowel following infections targeting the gastrointestinal tract. So, the investigators ought to know whether VS002A will be superior or not to WHO-ORS in the treatment of acute non-cholera watery diarrhea in infants and young children.

Hypothesis (if any): The amino acid-based ORS "VS002A" will reduce duration of non-cholera watery diarrhea in infants and young children when compared to treatment with standard WHO-ORS.

Objectives: To compare the efficacy of amino acid-based ORS "VS002A" compared to standard Glucose-based WHO ORS in infants and young children suffering from acute non-cholera watery diarrhea.

Methods:

* It will be a randomized, double-blind, two cell clinical trial at Dhaka Hospital of icddr,b. Total 312 (156 in each arm) male children aged 6-36 months old with acute (onset <48 hours) non-bloody watery diarrhea will be included in this study. However, patients with severe malnutrition, any systemic illness, cholera, unwilling to comply with study protocol, remain significantly dehydrated 4 hours after intravenous fluid infusion (if required at start), has documentation of taking antibiotics or antidiarrheal 48 hours before admission will be excluded.
* Intervention arm participants will get amino acid ORS (VS002A) and control arm will get standard glucose based WHO-ORS. Other aspects of clinical managements for diarrhea as per hospital guideline will be similar in both cases and controls

DETAILED DESCRIPTION:
Hypothesis to be tested:

The amino acid-based ORS "VS002A" will reduce the duration of non-cholera, watery diarrhea in infants and young children when compared to treatment with standard WHO-ORS.

Specific Objectives:

1. To evaluate and compare clinical responses (duration of diarrhea, stool output, ORS intake, and clinical success) in infants and young children suffering from acute non-cholera watery diarrhea treated with standard Glucose-based WHO ORS and amino acid-based ORS "VS002A".
2. To evaluate and compare electrolyte imbalance as possible complications in infants and young children suffering from acute non-cholera watery diarrhea treated with standard Glucose-based WHO ORS and amino acid-based ORS "VS002A".

Background of the Project including Preliminary Observations:

Diarrheal disorders constitute a leading cause of morbidity and mortality globally, and continue to be a major concern particularly for developing countries (Platts-Mills, 2015; WHO/UNICEF, 2013;Bern, 1992). Estimates show that in the year 2010, globally there were 1.7 billion episodes of diarrhea and 7.6 million deaths in children less than 5 years of age, mostly in the developing world; 72% of the deaths occurred in the first 2 years of life (Liu, 2012, 2015; Walker, 2013). In the Southeast Asian region, diarrhea is responsible for more than 20% of the total deaths among infants and young children (Liu, 2012, 2015).

Acute infectious diarrheal diseases are caused by a number of microbial pathogens. The bacterial pathogens include Vibrio cholerae, enterotoxigenic Escherichia coli, Shigella, Salmonella, and Campylobacter. Rotavirus is the most prominent viral diarrheagenic pathogen and also the leading cause of infantile diarrhea, whereas Entamoeba histolytica, Giardia lamblia and Cryptosporidia are the important parasites causing diarrhea. Based upon the pathogenetic mechanisms, these organisms may be broadly divided into two groups - secretory and invasive. V. cholerae is the prototype pathogen causing secretory diarrhea through liberation of an enterotoxin which stimulates intestinal secretion via intracellular accumulation of cyclic AMP (Fasano, 2002). There is insignificant inflammation or structural change in the intestinal mucosa and the diarrhea is watery in nature. Sufficient loss of fluids and electrolytes leads to dehydration, and thus the mainstay of treatment of patients with acute infectious secretory diarrhea is fluid replacement. On the other hand, Shigella (the prototype invasive pathogen) invades the gut mucosa and induces an inflammatory reaction, producing a dysenteric illness (Levine, 1982). The amount of fluid loss is minimal, and antibiotics are generally required in their management. In the developing countries, recent studies show that the commonest attributable microbial causes of moderate-to-severe diarrheal illnesses in infants and young children are: rotavirus, Cryptosporidium, enterotoxigenic E. coli producing heat-stable toxin (ST-ETEC, with or without co-expression of heat-labile enetrotoxin), and Shigella (Kotloff, 2013; Liu, 2016).

The standard clinical intervention in acute watery diarrhea is the use of oral rehydration solution (ORS), continued feeding, and oral zinc supplementation (WHO/UNICEF, 2013; WHO, 1995). The development of ORS for the treatment of dehydration due to diarrhea is one of the most significant therapeutic advances in the history of medicine. It is based upon the observations that even in a secreting small intestine it is possible to achieve a positive gut balance of fluid and electrolytes by adding glucose to the salt solution (Pierce, 1968; Fordtran, 1975). ORT is now recognized as a major scientific advance of utmost practical importance. The ORT solution currently recommended by the WHO/UNICEF contains glucose, sodium chloride, potassium chloride, and trisodium citrate dehydrate, which is optimal for rehydration of patients of all ages with dehydration from acute diarrhea of any etiology. It is estimated that ORS alone can successfully rehydrate 90% of patients with dehydration from acute diarrhea who previously would have required intravenous therapy therapy (Hirschorn, 1991).

However, ORT with the present ORS formulation has certain limitations - it does not reduce the volume, frequency or the duration of diarrhea (Mahalanabis, 1996). This is a constraint on the acceptance of ORT as a treatment of diarrhea, since the mothers and the health-care providers expect earlier recovery and a reduced severity of the disease, which is partly responsible for the widespread use of ineffective (and often harmful) antibiotics and other anti-diarrheal agents. These limitations prompted the development of the concept of improved ORS (initially termed 'super ORS') (Mahalanabis, 1986). Conceptually, an improved ORS should be able to reduce stool volume (by enhancing better reabsorption of fluid secreted into the small intestine), shorten duration of diarrhea (by reducing ileal effluent flow and stimulating colonic salvage), and reduce failure rate of ORT in patients with high purging rate. Several strategies were used to develop and test improved ORS - including the use of amino acids in addition to glucose, replacing glucose with glucose-polymers, using cereals instead of glucose, adding non-absorbable fermentable products to the ORS, and making the ORS hypo-osmolar by reducing both glucose and sodium concentrations. The recently recommended hypo-osmolar ORS is the result of intense search for such an improved ORS. Though the new hypo-osmolar ORS is more efficacious than the previously standard ORS, the duration of diarrhea is still not shortened, and there are failures with ORT (Alam, 1999). Thus, there is scope for further improvements of ORT.

The ORS takes advantage of the glucose-coupled intestinal sodium transport mechanism across the luminal membrane by the protein sodium glucose co-transporter 1 (SGLT1). Although nutrient independent sodium absorption across the intestinal epithelial brush border membrane is impaired in diarrhea, co-transport of sodium and glucose is preserved. This allows absorption of sodium and thus water as provided by oral rehydration solutions (Figure 1). Key in the success of use of ORS for rehydration is the fact that these physiological processes stay intact, even in the setting of severe diarrhea.

However, although ORS substantially enhances glucose-stimulated sodium absorption and correction of dehydration, it does not significantly decrease stool output, which is one of the main reasons for underutilization of ORS (Greenough, 1993; Wagner, 2015). Although an adequate explanation for this has not been established, it could be explained if glucose also stimulated anion secretion. In fact, based upon in vitro studies on the effect of glucose on active chloride and fluid secretion in mouse small intestinal cells and human colorectal adenocarcinoma (Caco-2) cells, glucose not only enhanced sodium absorption via SGLT1, a well-established phenomenon, but also stimulated active electrogenic chloride secretion via an increase in intracellular Ca2+ (Yin, 2014, AJP Cell). In clinical or experimental conditions, glucose-stimulated chloride secretion is most likely to occur in the villous cell region. These observations raise the possibility that in those clinical conditions in which there is villous damage and impaired glucose-stimulated sodium absorption, glucose may have deleterious effects on overall fluid and electrolyte movement by virtue of its stimulation of active chloride secretion.

In young children with acute non-cholera watery diarrhea, the rate of treatment failure due to clinically evident glucose intolerance is generally expected to be around 2% (Santosham M, 1982). However, 30% of young Peruvian children with acute diarrhea had detectable glucose malabsorption leading to treatment failure in 7% of the patients (Salazar-Lindo E, 1986). Thus, it may be hypothesized that simple dietary modifications and/or changes in the ORS formulation, such that glucose is replaced with compounds that do not stimulate chloride secretion, could significantly alter the outcome of the disease process.

Since certain neutral amino acids (e.g. glycine, L-alanine, L-glutamine) are also able to enhance the absorption of sodium ions and water, one approach to developing an improved ORS formulation was based on adding neutral amino acids or their dipeptides to WHO-ORS (Mahalanabis, 1983). The first studies of glycine-containing ORS were inconclusive; a meta-analysis of seven clinical trials conducted later showed that the ORS formulations containing glucose (or maltodextrin) and glycine (or glycyl-glycine) were not clinically superior to the standard WHO-ORS (International Study Group on Improved ORS, 1991). A summary of the eight clinical trials comparing L-alanine containing ORS with the WHO-ORS also showed variable results; in general, the differences in children with non-cholera diarrhea were not statistically significant (Bhan, 1994). Three clinical trials comparing glutamine-containing ORS with the WHO-ORS showed that it does not have any clinical advantage in children with non-cholera diarrhea (Bhan, 1994). One common thing among all the trials is that all the experimental amino acid-containing ORSs also contained glucose in variable amounts (9 g/L to 20 g/L); also most of these solutions had relatively high osmolarity (320 - 400 mosmol/L). One study which compared glucose-free glutamine-containing ORS with the WHO-ORS showed similar efficacy in children with acute non-cholera diarrhea (Gutierrez, 2007); it is to be noted that glutamine behaves like glucose in stimulating anion secretion (Yin, 2014). In a study comparing L-isoleucine supplemented glucose-containing ORS with WHO-ORS in young children with acute diarrhea, the differences were not statistically significant (Alam, 2011). However, in adult patients suffering from severe cholera, L-histidine-supplemented ORS was found superior to a histidine-free ORS; both the experimental and control solutions were rice-based and glucose-free (Rabbani GH, 2005). In another study, a glucose-free peptilose-based ORS was found more advantageous and acceptable than the WHO-ORS for treatment of mostly acute watery diarrhea among children (Simakachorn, 1993).

Previous studies on VS002:

Entrinsic Bioscience, a small business formed from intellectual property from the University of Florida (UF), developed a sugar-free, shelf-stable amino acid-based hydration medicinal food that effectively rehydrates, and improves barrier function of the bowel following infections targeting the gastrointestinal tract (GI). VS002's proprietary formulation of select amino acids contains no glucose. Studies in humans and animals demonstrate that sugar-free VS002 is an effective rehydration solution in a variety of circumstances.

Irradiation increases paracellular permeability in the gut with associated nutrient malabsorption, fluid imbalance, and bacterial translocation. In addition, irradiation induces active chloride ion secretion and fluid loss, and reduces transport of many carbohydrates, proteins and electrolytes. In a series of studies with radiation-induced enteritis with associated villus atrophy, an optimal composition of a novel ORS was defined based upon the observations that the inclusion of specific amino acids caused tightening of the mucosal barrier and reversal of symptoms of radiation-induced enteric dysfunction (Yin, 2014). VS002 thus consists of only the amino acids that improve electrolyte and water absorption and correct the increased gut permeability noted following irradiation and infectious disease.

It has been observed that certain amino acid-based pathways for sodium transport become the dominant pathway to compensate during times of stress. These pathways can be utilized to rehydrate the intestinal epithelial cells and restore normal bowel function. Eight specific amino acids retained their absorptive capacity from the gut lumen following radiation and at the same time decreased paracellular permeability: Lysine, Aspartic acid, Glycine, Isoleucine, Threonine, Tyrosine, Valine, and Serine.

Studies with VS002 have shown that VS002 administration i) rapidly rehydrates to increase fluid and electrolyte absorption, ii) tightens the mucosal barrier, thus decreasing local and systemic inflammation, and iii) increases crypt count and villus height, leading to an increase in the surface area of absorption. There is no toxicity associated with VS002 administration and the results of studies in animals and humans suggest that VS002 can serve as a highly safe and effective supportive care in place of standard ORS (Yin, 2014; Cheuvront, 2018; Clarke, 2018; Sollanek, 2018).

Results of In Vivo Studies Irradiated mice: Irradiated mice were treated either with saline or with VS002 for 14 days. Treatment with VS002 reduced mortality, preserved body weight, decreased pica (indication of nausea), and improved electrolyte and nutrient absorption (Yin, 2014; 2017) Mice with Rotavirus enterotoxin: Mice were exposed to rotavirus enterotoxin (NSP4) and sections of gut were tested for transport in vitro, and glucose-coupled sodium transport was found significantly impaired along with increased chloride secretion in the presence of NSP4. Glucose in the presence of NSP4 further increased the chloride secretion (Yin, 2017) Healthy Humans: Trials in healthy humans demonstrated i) VS002 safety; and ii) rehydration efficacy compared to a variety of commercial, glucose-containing beverages (sports drink, ORS). These studies included adults with diarrhea, healthy soldiers, young college students, and older adults (> 60 years old). Thus, administration of VS002 using eight amino acids to increase intestinal water and electrolyte absorption was associated with safe rehydration. See below for further study details.

VS002 was provided to > 250 adults treated for diarrhea in Indonesia and the Philippines. The consumption of VS002 was well tolerated by all subjects, with no adverse events (Olveda, 2016; Abdulah, 2018).

A study in healthy U.S. Soldiers and civilians (n = 26, males and females) examined the effect of rehydration via a common sports drink or VS002 after a bout of hypertonic or isotonic dehydration (3-4% body mass). Rehydration via VS002 resulted in improved rehydration of the extracellular space compared to the common sports drink, as well as greater fluid retention in the VS002 group (p < 0.05). The consumption of VS002 was well tolerated by all subjects, with no adverse events (Cheuvront, 2018).

Another study evaluated the ability of VS002 to optimize hydration compared to water in healthy adults (n = 40, males and females). Consumption of VS002 resulted in improved retention compared to water (p < 0.05). The consumption of VS002 was well tolerated by all subjects, with no adverse events (Sollanek, 2018).

The ability of VS002 to optimize hydration was also compared in younger and older adults (n = 24, males and females). Consumption of VS002 resulted in improved retention compared to water (p < 0.05). The consumption of VS002 was well tolerated by all subjects, with no adverse events (Clarke, 2019).

In a randomized, double-blind study to evaluate the efficacy of VS002, 587 adult patients received either WHO-ORS or VS002 to treat diarrhea. Safety results revealed that no patient consuming VS002 experienced any serious adverse events, whereas a small number of patients taking WHO-ORS did. Efficacy data for clinical cure rates were not clinically or statistically significant between treatment groups.

Therefore, it is hypothesized that VS002 will also be superior to WHO-ORS in the treatment of acute watery non-cholera diarrhea in infants and young children.

Advanced Amino acid-based ORS: VS002A Traditional oral rehydration solutions (ORS) contain sugars which stimulate intestinal sodium and water absorption through a variety of mechanisms. However, it has been under-appreciated that traditional ORS possess no anti-diarrheal functions and may exacerbate infectious diarrheal secretions (Yin et al., 2017).

Safety data of Advanced amino acid based ORS: VS002A

The food additive amino acids may be safely used as nutrients added to foods as individual amino acids in the free, hydrated, or anhydrous form, or as the hydrochloride, sodium, or potassium salts:

(1) L-Alanine; (2) L-Arginine; (3) L-Asparagine; (4) L-Aspartic acid; (5) L-Cysteine; (6) L-Cystine; (7) L-Glutamic acid; (8) L-Glutamine; (9) Aminoacetic acid (glycine); (10) L-Histidine; (11) LIsoleucine; (12) L-Leucine; (13) L-Lysine; (14) DL-Methionine (not for infant foods); (15) LMethionine; (16) L-Phenylalanine; (17) L-Proline; (18) L-Serine; (19) L-Threonine; (20) LTryptophan; (21) L-Tyrosine; (22) L-Valine.

EBS amino acid formulas are fully compliant with FDA 21 CFR requirements.

Gut health biomarkers Although oral rehydration therapy has greatly reduced diarrhoea-associated mortality, burden of diarrheal disease still persists in children below 5 years who are living under unsanitary condition and limited public health resources. This contributes to 43% of stunted growth and impaired cognitive development, affecting one-fifth of children worldwide and one-third of children in low- and middle-income countries (LMICs) (Guerrant, 2013; Kosek, 2013). Vicious cycle of enteric infection and malnutrition often leads to enteropathy for extended periods of time in young children when adequate water and sanitation are lacking (Guerrant, 2013; Owino, 2016). This type of enteropathy is known as Environmental Enteric Dysfunction (EED).

EED, previously known as tropical enteropathy or environmental enteropathy, is a sub-acute inflammatory condition of the small intestinal mucosa of unknown etiology (Ramakrishna, 2006). It is characterized by structural changes in the small intestine including villous atrophy and crypt hyperplasia compromising nutrient absorption and pathogenic barrier (increased permeability and inflammatory cell), impaired gut immune function, malabsorption, growth faltering, and generally asymptomatic, as distinct from diarrheal disease (Owino, 2016; Sullivan, 1991).

Data are limited from LMICs including Bangladesh on inflammatory and pathological changes in the gut wall like EED among children with diarrhea. In this study we will study plasma Citrulline (CIT) concentration as potential marker of functional enterocyte mass and absorptive functions of intestine, and Tryptophan-Kyanurenine (KT) ratio as a marker of gut inflammation.

CIT is an amino acid produced by intestinal epithelial cells and found lower in patients with enteropathy. One animal study reported lower plasma CIT level in the neonatal calves with diarrhea compared to healthy control (Gultekin, 2019). Tryptophan (TRP), a plant-derived essential amino acid (EAA) is needed to support growth and health in humans. In response to infection, TRP is mostly catabolized by an enzyme indoleamine 2,3-dioxygenase (IDO) to a toxic metabolite kynurenine (KYN). Low plasma TRP, high KYN and elevated KT ratio are found to be associated with infections (e.g. patients with inflammatory bowel disease suffer from diarrhoea) and chronic immune activation (Kosek, 2016).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6 months - 36 months,
2. Duration of diarrhea ≤48 hours,
3. Some dehydration (judged clinically according to the "Dhaka method"),
4. Written informed consent by either parent/guardian.

Exclusion Criteria:

1. Severe malnutrition (Weight-for-length WLZ/WHZ/WAZ <-3 or presence of nutritional edema)
2. Patients with diarrhea due to cholera.
3. Systemic illness (e.g. Pneumonia, tuberculosis, enteric fever, meningitis etc.)
4. Bloody diarrhea
5. Any congenital anomaly or disorder (e.g. diagnosed inborn error of metabolism, congenital cardiac disease, seizure disorders, hypothyroidism, Down's syndrome etc.)
6. Requirement of additional intravenous fluids after being provided with an IV for 4 hours on admission if severely dehydrated
7. Has documentation of taking antibiotic and/or antidiarrheal within the last 48 hours prior to hospitalization.

Ages: 6 Months to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — only male children, since separation of stool and urine is difficult in female children.
Enrollment: 312 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | upto 5 days after randomization
  Duration of diarrhea after randomization during hospital stay in hours

SECONDARY OUTCOMES:
Stool output | 1st 24 hours
  Stool output in the 1st 24 hours of hospitalization (g/kg body wt.), divided into two 12-hour periods
ORS intake | 1st 24 hours
  ORS intake in the 1st 24 hours of hospitalization (g/kg body wt.)

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No